CLINICAL TRIAL: NCT01159509
Title: The Effect of Hypertrophic Pyloric Stenosis (HPS) on Sodium Intake in Childhood
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: University of Haifa (Other)
Responsible Party: Dr. Ayala Maayan, Sheba Medical Center
Other Study IDs: SHEBA-10-8021-AM-CTIL
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Healthy; Hypertrophic Pyloric Stenosis
Keywords: hypertrophic pyloric stenosis; sodium intake; Healthy children with no chronic diseases; Status post HPS
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants ages -13 years that had HPS in infancy
  Interventions: Behavioral: sodium taste tests

INTERVENTIONS:
Behavioral: sodium taste tests — The cohort group will had sodium taste tests and an interview regarding diat habits.

SUMMARY:
The loss of sodium during infancy causes long term changes in sodium intake. Human research shows that the loss of maternal sodium during pregnancy and neonatal after birth causes an increase sodium intake during childhood. A study that examined sodium intake among infants that were treated with diuretics during the post-natal period found changes in sodium intake compared to controls. In this study we will test sodium intake in young children who have suffered from vomiting due to Hypertrophic Pyloric stenosis during early infancy.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-13 years
* Status post HPS in infancy

Exclusion Criteria:

* Children with chronic diseases
* Hospitalization due to dehydration after HPS hospitalization

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children ages 7-13 years. Status post HPS in infancy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Increased sodium intake | 1 year